CLINICAL TRIAL: NCT05335733
Title: Evaluation of Dental Plaque and Saliva Microbiome and Their Association With Periodontal Parameters in Premenopausal and Postmenopausal Women
Brief Title: Menopause and Oral Microbiome
Status: Completed | Type: Observational
Sponsor: Ege University (Other)
Collaborators: The Forsyth Institute (Other)
Responsible Party: Principal Investigator, Gülnur Emingil, Prof. Dr., Ege University
Other Study IDs: EGE BAP-23832
Record Dates: First submitted 2022-03-24; First posted 2022-04-19 (Actual); Last update posted 2024-01-02 (Actual); Status verified 2023-12

CONDITIONS: Menopause

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Postmenopausal women
  Interventions: Diagnostic Test: Intraoral examination, saliva, dental plaque and serum collection.
- Premenopausal women
  Interventions: Diagnostic Test: Intraoral examination, saliva, dental plaque and serum collection.

INTERVENTIONS:
Diagnostic Test: Intraoral examination, saliva, dental plaque and serum collection. — Probing pocket depth will be defined as the distance in millimeters from the gingival margin to the base of the gingival sulcus measured using a manual probe (Michigan 0 probe with Williams Markings) in all the teeth present except for third molars. Similarly, clinical attachment level (CAL) will be measured as distance from cementoenamel junction to the base of pocket and will be recorded manually to the nearest millimeter marking on probe.
  1 mililiter of saliva will be obtained by each participant. Subgingival dental plaque will be collected with sterile endodontic paperpoints from mesial sides of each natural teeth without a prostethic restoration. Serum samples will be also collected at the time of visit.

SUMMARY:
The study examines the saliva and dental plaque microbiome of women aged 35-65 in two groups: postmenopausal (case) and premenopausal (control). For this purpose, Illumina Platform to sequence 16S rRNA gene regions will be used. The data will be analyzed using the QIIME2 bioinformatics tool. Serum estradiol levels will be determined by the ELISA method. The investigators will examine the relationship between microbiome data (alpha diversity, beta diversity, and relative abundance) and menopausal status, estradiol levels, and periodontal health status using linear statistical models. Clinical samples of the study will be collected at Ege University, and the laboratory studies and sequence analysis will be conducted at the Forsyth Institute in Boston.

To obtain longitudinal data besides the cross-sectional data, the investigators will contact the participants of a previous study from 2019, whose saliva, dental plaque, and serum samples are currently being stored at -80 °C, and ask them to participate for a second sampling.

ELIGIBILITY:
Inclusion Criteria Regularly mensturating women over 35 years of age Postmenopausal women under 65 years of age

-

Exclusion Criteria:

- Antibiotic useage in last 3 months Being in menopausal transition phase

Ages: 35 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Middle aged women.
Sampling Method: Probability Sample
Enrollment: 220 (Actual)
Dates: Start 2022-02-15 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2023-10-30 (Actual)

PRIMARY OUTCOMES:
Differences in the relative abundances of bacteria in groups, acquired by processing of Illumina sequencing data with QIIME2 bioinformatic tool. | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Ege University, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided